CLINICAL TRIAL: NCT06908317
Title: Backward Chaining Method for Teaching the Getting Up From the Floor Among Long-Term Care Facility Residents
Brief Title: Teaching the Getting Up From the Floor Among Long-Term Care Facility Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Kovács Éva, college professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SE RKEB: 24/2025
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mobility Difficulty; Exercise; ELDERLY PEOPLE
Keywords: get up from the floor; backward chaining method; fall prevention; long-term care facility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Practicing in getting up from the floor is taught with backward chaning method, three times per week for 7 weeks plus usual care provided at the nursing home.
  Interventions: Other: floor rise training using backward chaining method
- usual care group (No Intervention): Practicing in only usual care

INTERVENTIONS:
Other: floor rise training using backward chaining method — Each session lasts for 40 minutes starting with a five minutes warming-up including flexibility exercises and ends with a five minutes cooling-down consisting of stretching and breathing exercises. Warming-up is followed by the practicing of getting up floor taught with BMC involving the following 7 steps:
  Step 1: descending from a standing position to half kneeling on a wedge pillow. Step 2: descending from a standing position to half kneeling on the floor. Step 3: Like step 2, then descending both knees to the floor into a high kneeling position. Step 4: Like step 3, then descending both hands to the floor one at a time, to come to a prone kneeling position. Step 5: Like step 4, then descending of the body to half sitting. A pillow can be positioned under the hip to soften the floor surface. Step 6: Like step 5, then descending of the body to side lying position. Step 7: Like step 6, then turning from side-lying to supine
  Arms: intervention group

SUMMARY:
The aim of this study is to determine the effect of teaching the getting up from the floor using the Backward Chaining Method on functional mobility, muscle strength, fear of falling, and life-space mobility among among long-term care facility residents.

Methods: Randomized controlled trial of a teaching the getting up from the floor using the Backward Chaining Method for older people living in long-term care facility. The assessment of primary and secondary outcomes takes place in all subjects upon entry to the study (pre-test) by blinded assessors and after the 20-session intervention (post-test). After baseline assessments is completed, participants will be randomly allocated to intervention or control groups using stratified randomization based on the use of walking aids and baseline values of FES-I.

The BCM sessions will be provided in a community room situated in the nursing home and will be led by a physiotherapist with extensive experience in geriatric physiotherapy with assistance of 2 physiotherapist student.

Only stable chairs provided for supporting and safety, wedge pillows, and training mats are required during practicing.

Expected results Improvement in functional mobility of the IG Improvement in lower and upper limb muscle strength Improvement in fall efficacy Improvement in life-space mobility

ELIGIBILITY:
Inclusion Criteria:

* • aged 65 years or older,

  * living in the nursing home for at least 2 months,
  * being able to walk at least 6 meters with or without walking aids

Exclusion Criteria:

* • being physically unable to be taught how to get up from the floor.

  * lower limb endoprosthesis implanted within 6 months
  * severe pain (VAS> 7/10)
  * cognitively unable to co-operate (based on psychiatrist's judgement)
  * planned moving away from the nursing home during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | Baseline and at the end of the 7-week intervention period
  A test to measure the time (in seconds) it takes for the participant to stand up from a standard armchair (approximate seat height 46 cm; arm height 65 cm), walk to a cone 3 m from the chair, turn around, walk back to the chair and sit down again. Instruction for the participants is given as follows "walk at a comfortable and safe pace". Wearing their usual footwear, using their usual walking aids, and supporting themselves on the arm of a chair to stand up are allowed/permitted, but physically assistance is not given for them.
  After a trial to familiarise the test, two successive performances are measured and the average of these is used the analyses. If necessary, a 30-second rest is provided between tests.

SECONDARY OUTCOMES:
30-second Sit to Stand Test | Baseline and at the end of the 7-week intervention period
  A test to assess the functional lower limb muscle strength. This test counts the sit-to-stands completed in 30 seconds by the participant from a chair (approximate seat height of 46 cm), with arms folded across the chest. The instruction to the participants is to " stand-up completely and sit down as quickly as possible". The digital stop-watch is started when begin on the command "go". Before timing, the participants is asked to perform one sit-to-stand. During testing, the completion of each correct stand is silently counted by the assessor to ensure for the participant his/her own correct performance. Incorrectly executed stands are not counted. At the end of 30-second test period, stand more than halfway up is counted as a full stand. If the participant could not perform a single sit-to-stand in a standard way, they are scored 0. During testing participants wear their regular footwear.
grip-strength | Baseline and at the end of the 7-week intervention period
  A test to assess overall muscle strength because this test strongly correlates with the overall muscle strength. The grip-strength will be measured by Kern MAP 40K1 dynamometer and measured in kilogram. This test will be administered in a sitting position and by taking the average of two consecutive measures in the dominant hand
Fall Efficacy Scale-International (FES-I) | Baseline and at the end of the 7-week intervention period
  A test to assess fear of falling. With its seven items, this scale asks how concerned the elderly person is about a possible fall during frequent activities of daily living. The answer is marked on a scale of four: 1=not at all concerned; 2=somewhat concerned; 3=fairly concerned; 4=very concerned. The total score can vary from 7 to 28 points with higher score indicating higher level of concern for falling
Nursing Home Life-Space Diameter (NHLSD) | Baseline and at the end of the 7-week intervention period
  A test to assess life-space mobility. It will be completed with the assistance of the nursing home staff based on the resident's movement during the previous 2 weeks. This measurement evaluates the extent of the resident's movement (diameter): (1) within resident's room, (2) within unit, (3) outside unit, and (4) outside the facility; and frequency of movement: (0) never, (1) less than weekly, (2) at least weekly, (3) > 2 times/week, (4) 1-3 times/day, and (5) > 3 times/ day. Total NHLSD scores were calculated as 1(diameter 1 × frequency 1) + 2(diameter 2 × frequency 2) + 3(diameter 3 × frequency 3) + 4(diameter 4 × frequency 4). The score ranges from 0 to 50, 0 indicating being bedbound and 50 indicating leaving the facility daily. The total scores marks the area in which the person moves around. The total score ranges from 0 to 50, 0 indicating being bedbound and 50 indicating leaving the facility daily
independence of mobility | Baseline and at the end of the 7-week intervention period
  During using the Nursing Home Life-Space Diameter (NHLSD), besides distance and frequency, the human assistance for mobility is scored on a two-point scale (0 = dependent, 1 = independent). If movement is performed without human assistance, score of each item is multiplyed by 2. This another total score incorporates mobility independence into the total score and thus reflects not only distance and frequency but also dependence on human assistance for mobility. In this case the maximum score, NHLSD-dependence, is 100 points
Number of falling | During the 7-week intervention period
  Falls will be recorded to measure adverse events. It will be by nursing home staff throughout the intervention period. They will be provided with a pre-designed diary and asked to record each day if any participants will have fallen. The diaries will be collected weekly by the assessor physiotherapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.